CLINICAL TRIAL: NCT05761405
Title: Metabolic Potentiation of Aminoglycosides: a Novel Antimicrobial Strategy to Prevent Urinary Tract Infections (UROPOT TRIAL).
Brief Title: Potentiated Aminoglycosides in Postoperative Urinary Tract Infection Prophylaxis
Acronym: UROPOT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Sylvain Meylan, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-001979
Record Dates: First submitted 2022-11-15; First posted 2023-03-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections; Urological System Complication of Procedure
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ceftriaxone; Amikacin

STUDY DESIGN:
Intervention Model Description: Randomized, multicentre, double-blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pharmacy prepares a randomization list with an additional 20% to account for drop-outs. Based on this, the pharmacy prepares labels (study ID, local center ID, subject ID) and a randomization list (subject ID, open-label treatment (i.e. AMK, AMK+MAN, CRO)). These are delivered to the blinded to the patient awaiting surgery with anonymized subject IDs (consecutive numbering). The investigator has no access to this list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ceftriaxone (CRO) (Active Comparator): Ceftriaxone infusion. Ceftriaxone is a beta-lactam antibiotic that is the standard-of-care antibiotic for prophylaxis of asymptomatic bacteriuria in Switzerland. The choice of 2000 mg delivered intravenously reflects the general practice.
  Interventions: Drug: Ceftriaxon
- Aminoglycoside (AMK) (Active Comparator): Amikacin infusion Amikacin is an aminoglycoside routinely used in Australia (e.g. amikacin, gentamicin) as the standard of care for antibiotic prophylaxis for endourological treatments. It is also used globally for fever in neutropenia in hematological patients. Due to their relatively limited use, aminoglycosides have low resistance rates amongst Enterobacteriaceae. A single dose of 1000mg will be used intravenously
  Interventions: Drug: Amikacin
- AminoglycosideLD + Mannitol (AMK1/2 + MAN) (Experimental): Amikacin + Mannitol combination The addition of Mannitol enhances bactericidal effect of amikacin in E.coli and K.pneumoniae in animal models and allows for a decrease of amikacin dosing. A single dose of 500mg (low dose or LD - decrease by 50%) systemic amikacin will be used intravenously in combination with 5 grams mannitol delivered intravenously.
  Interventions: Combination Product: mannitol-enhanced aminoglycoside

INTERVENTIONS:
Combination Product: mannitol-enhanced aminoglycoside — Preselected patients with ureteral stents in situ who are scheduled to undergo endourological ureteral stent manipulation will have routine urine cultures prior to intervention.
  Procedures: Consented patients will be randomized for the type of antibiotic prophylaxis according to a global randomization list (i.e. CRO, AMK, AMK1/2+MAN)).
  Antibiotics (± mannitol) will be delivered in a single infusion that will be administered within 30 minutes.
  Arms: AminoglycosideLD + Mannitol (AMK1/2 + MAN)
Drug: Ceftriaxon — Preselected patients with ureteral stents in situ who are scheduled to undergo endourological ureteral stent manipulation will have routine urine cultures prior to intervention.
  Procedures: Consented patients will be randomized for the type of antibiotic prophylaxis according to a global randomization list (i.e. CRO, AMK, AMK1/2+MAN)).
  Antibiotics will be delivered in a single infusion that will be administered within 30 minutes.
  Arms: Ceftriaxone (CRO)
Drug: Amikacin — Preselected patients with ureteral stents in situ who are scheduled to undergo endourological ureteral stent manipulation will have routine urine cultures prior to intervention.
  Arms: Aminoglycoside (AMK)

SUMMARY:
Urinary tract hardware such as pig-tail catheters are are frequently used for management of urolithiasis or other obstructive pathologies. They are readily colonized by urogenital flora leading to asymptomatic bacteriuria. While asymptomatic bacteriuria is not per se a problem for patients, it may lead to severe infections in the context of hardware manipulation leading to mucosal damage (e.g. catheter exchanges or stone extraction). Such interventions therefore warrant an antibiotic prophylaxis. However, bacteria rapidly form biofilms on hardware; aside of fluoroquinolones, antibiotics have limited anti-biofilm activity. Furthermore, the widespread use of antibiotics has lead to resistant strains. Hence, novel antimicrobial strategies are needed. Recently, metabolism-based potentiation of aminoglycoside has shown high antimicrobial activity against persistent forms of bacteria such as biofilms in the context of murine catheter-associated urinary tract infections. Because of the highly favorable pharmacodynamic profile of aminoglycoside in the urinary tract and the metabolic potentiation, aminoglycosides can be reduced to levels with minimal toxicity.

UROPOT aims to compare the efficacy of potentiated aminoglycoside to standard of care for (i) prophylaxis of asymptomatic bacteriuria during urinary hardware manipulations with mucosal trauma (Pig-tail catheter exchange, stone surgery with prior in-dwelling catheter, etc.) and (ii) sustained microbiological eradication through antibiofilm activity. UROPOT will compare the rate of post-interventional urinary tract infections (primary outcome). It will also assess safety and eradication potency (microbiological outcome).

DETAILED DESCRIPTION:
UROPOT is a randomized, single-centre, double-blind, pilot trial comparing a combination of aminoglycosides and mannitol to standard of care or aminoglycosides alone for the peri-operative antimicrobial prophylaxis of endourological procedures with mucosal trauma in the presence of hardware. Adults (≥18 years) scheduled for such procedures with mucosal trauma (stone surgery with hardware, pig-tail catheter exchanges) and having an asymptomatic bacteriuria E. coli or K. pneumoniae as identified 10 days prior to surgery, will be randomly assigned (1:1:1) to receive standard prophylaxis (gen. Ceftriaxone 2 g) for 24 hours, a single dose of amikacin (6mg/kg i.v.) or a single dose of mannitol (pres. 2.5g i.v. bolus)/amikacin (3mg/kg i.v.). Sample size for the three groups will be constructed to demonstrate a non-inferiority for the clinical outcome (absence of infectious complication within 48 hours from operation) with a power of 80%. Complications in the absence of antimicrobial prophylaxis range from 2-10%. Patients will be excluded if baseline urine culture has another bacterial pathogen or E. coli or K. pneumoniae are documented to be aminoglycoside resistant. The primary endpoint will be the prevention of complications(clinical) that will be evaluated for non-inferiority compared to the accepted standard of care. i.e., within a 6% margin Assuming a rate of complication as low as 2%, the new treatments will be considered non-inferior if the corresponding rate of complication is not above 8% (i.e., 6% margin). This non-inferiority margin can be evaluated with a total for 128 patients per treatment arm, at 1-sided alpha of 5%, with power 80%, through an exact two-sample test for proportions. Two comparisons will be performed of arm A and of arm B versus standard of care (SoC). In addition, a microbiological outcome will be included to document higher biofilm eradication rate. This will be documented by sonication of extracted hardware as well as repeat urine culture at post-operative days 7 and 14 days (secondary outcomes). Safety will be monitored with a specific focus on nephrotoxicity and ototoxicity. If highly efficient, this novel antimicrobial strategy would be expanded to treatment of complicated urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adults (≥18 years)
* Ureteral stent in situ
* Patients scheduled for endourological ureteral manipulations (e.g. endourological stone surgery, ureteral stent exchange)
* Asymptomatic bacteriuria with strains of E. coli and/or K. pneumoniae sensitive to Ceftriaxone and Amikacin/Aminoglycosides.

Exclusion Criteria:

* Allergy to one of the study drugs Beta-lactams, aminoglycosides or mannitol
* Pregnant and lactating women
* Glomerular filtration rate (CKD-EPI eGFR) < 50ml/min / 1,73m2
* Hearing impairment
* Myasthenia gravis or other forms of myoneural disorders
* Congestive heart failure, Pulmonary edema
* Intracranial hemorrhage, blood-brain barrier compromise
* Previous (within 3 months prior to randomization) or concomitant participation in another interventional clinical trial
* Antibiotic treatment within 14 days prior to randomization
* Mixed cultures of E. coli and/or K. pneumonia with other bacteria
* Inability to understand and follow the protocol
* Inability to give informed consent
* BMI<20 or >30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Infection prophylaxis | 48 hours postoperatively
  Incidence of postoperative infections within the initial 48 hours postoperatively.

SECONDARY OUTCOMES:
Combined microbiological eradication | 6-8 hours post infusion
  anti-biofilm activity as determined by culture of sonicated catheter (CFU/ml) and intraoperative urine culture (CFU/ml)
Sustained microbiological eradication | Up to 2 weeks
  To document eradication of bacteriuria at postoperative day 2 and 14 day by urine culture (CFU/ml)
Surgical safety outcome | Day 0-14
  Postoperative complications
Pharmacokinetics outcome | Day 0, Day 2, Day 14
  Measurements of maximum urine drug concentrations (Amikacin, Ceftriaxone, Mannitol)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 0-Day 14
  Safety and tolerability of Amikacin/Mannitol combination (serious adverse events (SAEs), pre-specified adverse events (AEs) of special interest (ototoxicity, nephrotoxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Meylan, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Stritt K, Roth B, Masnada A, Hammann F, Jacot D, Domingos-Pereira S, Crettenand F, Bohner P, Sommer I, Breat E, Sauser J, Derre L, Haschke M, Collins JJ, McKinney J, Meylan S. UROPOT: study protocol for a randomized, double-blind phase I/II trial for metabolism-based potentiation of antimicrobial prophylaxis in the urological tract. Trials. 2024 Oct 15;25(1):682. doi: 10.1186/s13063-024-08526-7. PMID 39407325